CLINICAL TRIAL: NCT06702930
Title: The Effects of Morning vs. Evening High-intensity Interval Exercise on the Magnitude of the Morning Blood Pressure Surge
Brief Title: Exercise Timing on the Morning Blood Pressure Surge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Philip Millar, Associate Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 19-07-002
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Post-Exercise Hypotension; Ambulatory Blood Pressure Monitoring; High-intensity Interval Exercise
Keywords: Ambulatory blood pressure monitoring; Morning blood pressure surge; High-intensity interval exercise; Post-exercise hypotension
MeSH Terms: conditions — Post-Exercise Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No exercise was performed and ambulatory blood pressure was assessed for 24 hours.
- Morning high-intensity interval exercise (Experimental): High-intensity interval exercise was performed between 8-10 am and ambulatory blood pressure was assessed for 24 hours after.
  Interventions: Other: Morning high-intensity interval exercise
- Evening high-intensity interval exercise (Experimental): High-intensity interval exercise was performed between 5-7 pm and ambulatory blood pressure was assessed for 24 hours after.
  Interventions: Other: Evening high-intensity interval exercise

INTERVENTIONS:
Other: Morning high-intensity interval exercise — High-intensity interval exercise was performed between 8-10 am
  Arms: Morning high-intensity interval exercise
Other: Evening high-intensity interval exercise — High-intensity interval exercise was performed between 5-7 pm
  Arms: Evening high-intensity interval exercise

SUMMARY:
The goal of this clinical trial was to assess the effects of morning vs. evening high-intensity interval exercise on the magnitude of the morning blood pressure surge in young healthy adults. The main questions it aimed to answer were:

* Does the timing of high-intensity interval exercise modulate the magnitude of the morning blood pressure surge?
* Do sex differences exist?

Participants came in and completed a bout of high-intensity interval exercise in the morning (8-10 am) and evening (5-7 pm) as well as a no exercise control, and ambulatory blood pressure was assessed for 24 hours afterwards.

DETAILED DESCRIPTION:
Introductory Visit:

Participants came in for 4 visits. The first visit was an introductory visit where chronotype, eligibility for exercise, and anthropometrics were measured. This was followed by a maximal incremental exercise test to determine aerobic capacity (i.e., V̇O2peak) on a cycle ergometer, and instrumentation of an ambulatory blood pressure monitor for familiarization during daily activities and sleep.

Intervention Visits:

Three intervention visits (control, morning exercise, and evening exercise) were completed. The order was randomized using and each visit was separated by a minimum of 36 hours. Each intervention visit began by obtaining the participant's resting blood pressure and heart rate and ended with the instrumentation of the ambulatory blood pressure monitor. No exercise was performed during the control visit. The morning exercise visit included a bout of high-intensity interval exercise between 8-10 am and the evening exercise visit included a bout of high-intensity interval exercise between 5-7 pm. The high-intensity interval exercise protocol consisted of a light intensity, 3-minute warm-up at 15% peak power followed by ten 1-minute work intervals at 80% of peak power, with each interval separated by 1-minute rest intervals at 15% peak power. A 3-minute cool down was performed at 15% peak power.

ELIGIBILITY:
Inclusion:

* Between 18-50 years of age.
* No history of known disease.
* None smokers.
* No use of chronic medications other than oral contraceptives.

Exclusion:

* <18 years of age.
* >50 years of age.
* Cardiovascular disease.
* Metabolic disease.
* History of smoking (within the past 3 months).
* Chronic medications (other than oral contraceptives).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Morning blood pressure surge | Through study completion, an average of 4 weeks.
  The difference between morning blood pressure (the mean of the 4 blood pressure readings after awakening) and sleep-trough blood pressure (the mean of the lowest blood pressure during sleep and two adjacent blood pressure readings).

SECONDARY OUTCOMES:
Nighttime blood pressure dip | Through study completion, an average of 4 weeks.
  The percent difference between daytime blood pressure (average of all blood pressure readings when participants reported being awake) and nighttime blood pressure (average of all blood pressure readings when the participant reported being asleep).

CONTACTS AND LOCATIONS:
Overall Officials: Julian Bommarito, MSc, Study Director — University of Guelph; Philip Millar, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: After publication; unending.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Derived] Bommarito J, Millar PJ. The effects of morning versus evening high-intensity interval exercise on the magnitude of the morning blood pressure surge. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-11. doi: 10.1139/apnm-2024-0449. PMID 39689295